CLINICAL TRIAL: NCT02702141
Title: A Phase 1, Open-label, Dose-escalation Study of SGN-CD19B in Patients With Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphoma
Brief Title: A Safety Study of SGN-CD19B in Patients With B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN19B-001
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Non-Hodgkin Lymphoma; DLBCL; Diffuse Large B-cell Lymphoma; Grade 3 Follicular Lymphoma
Keywords: Non-hodgkin lymphoma; Antibody-drug conjugate; CD19; Diffuse large B-cell lymphoma; DLBCL; Grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — SGN-CD19B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGN-CD19B (Experimental)
  Interventions: Drug: SGN-CD19B

INTERVENTIONS:
Drug: SGN-CD19B — Given intravenously Day 1 of 28-day or 42-day cycles

SUMMARY:
The study will examine the safety profile of SGN-CD19B administered as a single agent. The main purpose of the study is to estimate the highest dose that does not cause unacceptable side effects of SGN-CD19B in patients with relapsed or refractory aggressive B-cell non-Hodgkin lymphoma (NHL) subtypes of diffuse large B-cell lymphoma (DLBCL) and Grade 3 follicular lymphoma (FL3). Additionally, the pharmacokinetic profile and antitumor activity of SGN-CD19B will be assessed.

DETAILED DESCRIPTION:
SGN-CD19B will be given to patients at increasing doses every 28 days (or on an alternative dosing schedule of every 42 days).

Individual expansion cohorts of up to approximately 20 patients will be opened at dose levels selected by the Safety Monitoring Committee based on the aggregate known safety and activity data to further define the safety and antitumor activity in refractory and relapsed disease subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed, refractory, or progressive disease following at least 2 prior systemic therapies
* Measurable disease
* Eastern Cooperative Oncology Group status of 0 or 1
* Adequate baseline renal and hepatic function

Exclusion Criteria:

* Prior treatment with CD19 directed agents unless CD19 expression is confirmed after completion of CD19-directed treatment
* Known HIV, active hepatitis B or active hepatitis C infection
* Prior allogeneic stem cell transplant
* Inadequate lung function
* Anticancer treatment within 4 weeks of study drug or 2 weeks if patient experienced disease progression on prior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose
Incidence of laboratory abnormalities | Through 1 month following last dose

SECONDARY OUTCOMES:
Blood concentrations of SGN-CD19B | Through 3 weeks after dosing
Incidence of antitherapeutic antibodies | Through 1 month following last dose
Objective response rate | Through 1 month following last dose
Rate of response | Through 1 month following last dose
Progression-free survival | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pinelli, PA-C, MMSc, Study Director — Seagen Inc.
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University (NYU) Cancer Institute, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, The, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Ryan MC, Palanca-Wessels MC, Schimpf B, Gordon KA, Kostner H, Meyer B, Yu C, Van Epps HA, Benjamin D. Therapeutic potential of SGN-CD19B, a PBD-based anti-CD19 drug conjugate, for treatment of B-cell malignancies. Blood. 2017 Nov 2;130(18):2018-2026. doi: 10.1182/blood-2017-04-779389. Epub 2017 Sep 13. PMID 28903943